CLINICAL TRIAL: NCT00507780
Title: Use of the GnRH Agonist Leuprolide Acetate (Lupron(Registered Trademark)) to Preserve Ovarian Function in Women Undergoing Chemotherapy
Brief Title: Effect of Cetrorelex Acetate on Ovarian Function in Women Undergoing Chemotherapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Alicia Y. Armstrong, M.D./National Institute of Child Health and Human Development, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 070193; 07-CH-0193
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-07-22

CONDITIONS: Ovarian Function; Preservation of Ovarian Function
Keywords: GnRH Antagonist; Premature Ovarian Failure; Fertility; Chemotherapy; POF
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

INTERVENTIONS:
Drug: GnRH antagonist

SUMMARY:
This study will examine whether the drug cetrorelex acetate (Cetrotide[Registed Trademark]) can protect ovarian function in women undergoing chemotherapy. Some cancer treatments are known to cause a change in women's periods or to cause menstruation to stop completely, so that they cannot become pregnant. Cetrorelex acetate has been used for many years to lower hormone levels and stop periods in patients undergoing in vitro fertilization treatments. This study will see if making the ovaries inactive may protect them from being affected by certain cancer drugs, and thus preserve fertility.

Women up to age 21who have begun menstruating, who have their uterus and at least one functioning ovary, and who are undergoing chemotherapy with cyclophosphamide, busulfan, nitrogen mustard or L-phenalanin mustard may be eligible for this study.

Participants undergo the following procedures during this 24-month study:

Baseline evaluation

* Medical history, physical examination and blood and urine tests
* Questionnaire about quality of life, menstrual periods, vaginal bleeding and desire for future fertility
* 3D ultrasound of abdomen
* DEXA scan to evaluate bone density

Assignment to treatment with:

* Lo ovral (contraceptive pill to prevent pregnancy and control menstrual periods) alone, or
* Lo ovral and the study drug cetrorelex acetate, given as an injection under the skin once a day for six menstrual cycles

Evaluations

* Transvaginal 3D ultrasound to monitor changes in the ovary - after 6 months of cetrorelex acetate injections
* DEXA scan - after 6 months of cetrorelex acetate injections
* Blood tests for safety monitoring, pregnancy testing, endocrine tests and research uses - every 3 months during first year, every 6 months during second year
* Questionnaire to monitor changes and quality of life - every 3 months during first year, every 6 months during second year.

DETAILED DESCRIPTION:
As a result of the inability of female germ cells to regenerate after injury, a number of chemotherapeutic agents induce premature ovarian failure in the majority of reproductive age women who receive them. The long-term survival for these women has increased with more effective chemotherapies, making iatrogenic ovarian failure and infertility an increasingly significant issue. Currently the choices for maintaining fertility include in vitro fertilization (IVF) and embryo cryopreservation, oocyte cryopreservation and the use of GnRH agonist and antagonist to preserve ovarian function.

Much of the evidence for the use of GnRH agonist to prevent premature ovarian failure is found in the systemic lupus erythematosus literature. Blumenfeld and colleagues have published a report that demonstrates preservation of ovarian function in 100% of patients treated with leuprolide acetate prior to cyclophosphamide therapy, compared to a 50% ovarian failure rate in patients not receiving leuprolide acetate. Although the results of animal studies and human studies are encouraging, adequately controlled trials are needed. Future trials will need to have sufficient numbers of patients, receiving multiple types of chemotherapeutic agents to adequately document the utility of medical prophylaxis. The experience with ovulation induction suggests GnRH antagonists may have similar efficacy to GnRH agonists. GnRH antagonists compete directly with GnRH in receptor binding, and as a result antagonists rapidly inhibit secretion of gonadotropin and sex steroids. Unlike GnRH agonists, GnRH antagonists have an immediate effect and antagonists can be given independent of menstrual cycle day. These differences represent several practical benefits offered by an antagonist. In a recent case series by Sauer et al, cetrorelix acetate, a GnRH antagonist, was given in doses of 3mg at four day intervals to four patients ages 21-30. Menses was preserved in all four patients and there was one spontaneous conception. Because of the potential advantages of the use of a GnRH antagonist when compared to an agonist, cetrorelix acetate will be studied against placebo in this investigation.

Our specific aim is to compare the rates of ovarian preservation in reproductive age women receiving chemotherapeutic agents known to affect ovarian function who receive Cetrorelix acetate co treatment with women who receive these agents and do not receive Cetrorelix acetate. A second aim is to evaluate the ability of the Cetrorelix acetate co treatment to induce therapeutic amenorrhea in a study population at risk for thrombocytopenia and associated heavy vaginal bleeding.

ELIGIBILITY:
* INCLUSION CRITERIA:

All reproductive age women menarche - age 21, undergoing chemotherapy with agents known to affect ovarian function that have a follicle stimulating hormone level (FSH) less than 20 mIU/L will be offered enrollment. We define premature ovarian failure as the development before age 40 years of greater than 4 months of amenorrhea or menstrual irregularity, associated with two serum FSH levels in the menopausal range (sampled at least 1 mo apart).

EXCLUSION CRITERIA:

FSH greater than 20 mIU/L

Sensitivity or allergy to oral contraceptives (lo ovral) or cetrorelix acetate

Patients who have had surgical removal of their ovaries

Patients who are currently pregnant or attempting conception

Severe renal impairment

Premenarchal patients

Patients greater than 21

Patients who have undergone radiation therapy or who are scheduled to undergo radiation therapy during the study period.

Patients with a family history of premature ovarian failure

Ages: 10 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07-18; Primary Completion 2010-07-22 (Actual); Study Completion 2010-07-22 (Actual)

PRIMARY OUTCOMES:
Antimullerian hormone, ovarian follicle count | 2-years

SECONDARY OUTCOMES:
Menstrual history | 2-years

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Oktay KH, Yih M. Preliminary experience with orthotopic and heterotopic transplantation of ovarian cortical strips. Semin Reprod Med. 2002 Feb;20(1):63-74. doi: 10.1055/s-2002-23520. PMID 11941536
- [Background] Donnez J, Dolmans MM, Demylle D, Jadoul P, Pirard C, Squifflet J, Martinez-Madrid B, van Langendonckt A. Livebirth after orthotopic transplantation of cryopreserved ovarian tissue. Lancet. 2004 Oct 16-22;364(9443):1405-10. doi: 10.1016/S0140-6736(04)17222-X. PMID 15488215
- [Background] Teinturier C, Hartmann O, Valteau-Couanet D, Benhamou E, Bougneres PF. Ovarian function after autologous bone marrow transplantation in childhood: high-dose busulfan is a major cause of ovarian failure. Bone Marrow Transplant. 1998 Nov;22(10):989-94. doi: 10.1038/sj.bmt.1701483. PMID 9849696